CLINICAL TRIAL: NCT02834884
Title: SPECTA: Screening Cancer Patients for Efficient Clinical Trial Access
Acronym: SPECTA
Status: Recruiting | Type: Observational
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC-1553
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: All Tumor Types
Keywords: rare cancer; biomarker; molecular screening; cancer; biobanking
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — FFPE tissue sample; Blood sample; Fresh bone marrow sample (in case of hematological malignancies)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- RP-1828 IMMUcan (CLOSED for recruitment since August 2024): The goal is to generate broad molecular and cellular profiling data of the tumour and its microenvironment from cancer patients integrated with clinical data, to understand how the immune system and tumours interact, and the impact of current therapeutic interventions.
  Tumor types: Thorax, Head and Neck, Breast, Gastrointestinal, Genito Urinary
  Interventions: Genetic: RP-1828 IMMUcan
- RP-1759 AYA/TYA (CLOSED for recruitment since December 2021): The pilot study will be focusing on young adults (12 to 29 years old) with rare cancer to understand better the biology of the tumor in this specific population, and compare it to children and adults with similar disease, as well as to improve the inclusion of young adults into clinical trials.
  Tumor type: CNS
  Interventions: Genetic: RP-1759 AYA/TYA
- RP-1843 Arcagen (CLOSED for recruitment since November 2022): This is a collaborative project between EORTC and EURACAN to perform molecular characterisation of rare cancers patients, using Foundation Medicine tests. The goal of this project is to get a better understanding of the genomic landscape of rare cancers and potentially help define possibilities for targeted treatments/clinical trials for this population.
  Tumor types: all 10 EURACAN domains
  Interventions: Genetic: RP-1843 Arcagen
- RP-1920 BioRadon: The primary objective is to assess the correlation between the molecular profiles of NSCLC patients and indoor radon concentration, measured with an alpha-particle detector (a standardized and validated way of measuring indoor radon).
  Tumor type: Thorax
  Interventions: Genetic: RP-1920 BioRadon

INTERVENTIONS:
Genetic: RP-1828 IMMUcan — WES, lcWGS and RNAseq, multiplex IF and IMC
  Groups: RP-1828 IMMUcan (CLOSED for recruitment since August 2024)
Genetic: RP-1759 AYA/TYA — WES, RNAseq and EPIC array
  Groups: RP-1759 AYA/TYA (CLOSED for recruitment since December 2021)
Genetic: RP-1843 Arcagen — NGS panel
  Groups: RP-1843 Arcagen (CLOSED for recruitment since November 2022)
Genetic: RP-1920 BioRadon — NGS panel
  Groups: RP-1920 BioRadon

SUMMARY:
SPECTA is a quality assured platform for collecting clinicopathologically annotated biological material, imaging data, operative images, environmental assessment, questionnaires as well as patient-reported outcomes from cancer patients to support biospecimen-based translational research and clinical cancer research, including biomarker discovery to improve the understanding of tumor biology and cancer patients care.

DETAILED DESCRIPTION:
Patients are recruited in the platform for the research purpose of 4 downstream projects. For more information, please have a look at the "Groups and cohorts" section.

ELIGIBILITY:
* Patients with pathologically confirmed selected tumor types (at site or centrally);
* Mandatory availability of adequate human biological material (HBM);
* Centrally performed confirmation of HBM adequacy in terms of quality and quantity for SPECTA downstream project requirements;
* Age ≥ 12 years;
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule;
* Written informed consent according to applicable legal and ethical requirements;

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pathologically confirmed selected tumor types.
Sampling Method: Non-Probability Sample
Enrollment: 4975 (Estimated)
Dates: Start 2017-05-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
To establish a quality assured platform to improve the understanding of tumor biology and cancer patients care | 5 years
  material (including imaging data) as well as patient-reported outcomes from patients with cancer diagnosis to support biospecimen-based translational research and biomarker discovery to improve the understanding of tumor biology and cancer patients care.

SECONDARY OUTCOMES:
To perform biospecimen and data based high quality research aiming to better understand the biology of cancer, and/or how it is currently managed and/or how to better diagnose and treat it in the future; | 5 years
To investigate the molecular pathways related to the development of specific tumors from a biological point of view; | 5 years
To investigate the effect of cancer treatment on the tumor, microenvironment and patients globally; | 5 years
To collect large series of homogeneous clinical data to analyse the disease course and treatment performed; | 5 years
To investigate the prevalence and validate the prognostic or predictive value of novel biomarkers in cancers; | 5 years
To perform biospecimen and data based high quality research aiming to facilitate the discovery of new test for tumor biomarkers or facilitate the establishment of validated tests for tumor biomarkers; | 5 years
To identify patients with molecular alterations in their tumor that can be matched to biomarker-driven clinical trials, to facilitate enrollment of cancer patients in biomarker-driven clinical trials. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Besse, Pr., Study Chair — European Organisation for Research and Treatment of Cancer - EORTC
Locations (134):
- Medical University Vienna - General Hospital AKH, Vienna, Austria
- Belgium (13):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - ZAS Middelheim, Antwerp
  - Hopitaux Universitaires - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Pole Hospitalier Jolimont - Hopital Jolimont, Haine-Saint-Paul
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
  - C.H.U. Sart-Tilman, Liège
  - Centre Hospitalier Regional De La Citadelle, Liège
  - CHU Site Sainte-Elisabeth-UCL Namur, Namur
  - AZ Turnhout - Campus Sint Elisabeth, Turnhout
  - CHU Mont Godinne - UCL Namur, Yvoir
- University Hospital Centre Zagreb, Zagreb, Croatia
- Bank Of Cyprus Oncology Centre, Stróvolos, Cyprus
- University Hospital Motol, Prague, Czechia
- North Estonia Medical Centre - Mustamäe unit, Tallinn, Estonia
- France (37):
  - Centre Hospitalier Avignon, Avignon
  - CHRU de Besancon - Hopital Jean Minjoz, Besançon
  - Centre de Radiotherapie Pierre Curie, Beuvry
  - CHU de Bordeaux - Groupe Hospitalier Saint-Andre - Hopital Saint-Andre, Bordeaux
  - Institut Bergonie, Bordeaux
  - Centre Hospitalier - Boulogne Sur Mer, Boulogne-sur-Mer
  - CHU de Lyon - Hopital Louis Pradel, Bron
  - CHU Lyon - Hopital neurologique Pierre Wertheimer, Bron
  - Centre Francois Baclesse, Caen
  - Centre Hopitalier Intercommunal De Creteil, Créteil
  - Centre Georges-Francois-Leclerc, Dijon
  - CHU de Grenoble - La Tronche - Hôpital A. Michallon, Grenoble
  - Centre Hospitalier Departemental Vendee, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - CHRU de Lille, Lille
  - CHU de Lyon - Hopital Edouard Herriot, Lyon
  - Centre Léon Berard, Lyon
  - CHU de Lyon - Hopital Lyon Sud, Lyon
  - Assistance Publique - Hopitaux de Marseille - Hopital Nord, Marseille
  - Centre Hospitalier D'Annecy Genevois, Metz-Tessy
  - CHU Montpellier-Hopital Arnaud De Villeneuve, Montpellier
  - Institut du Cancer de Montpellier, Montpellier
  - Centre Hospitalier Des Pays De Morlaix, Morlaix
  - Centre d'Oncologie de Gentilly, Nancy
  - CHU de Nice - Hopital De L'Archet, Nice
  - Assitance Publique - Hopitaux de Paris - Hopital Saint-Louis, Paris
  - Assistance Publique - Hopitaux de Paris - Hopital Saint Antoine, Paris
  - Assistance Publique - Hopitaux de Paris - La Pitie Salpetriere, Paris
  - Institut Curie- Hopital de Paris, Paris
  - Groupe Hospitalier Paris Saint-Joseph - Hopital Saint Joseph, Paris
  - Centre Eugene Marquis, Rennes
  - Institut de Cancerologie de l'Ouest (ICO) - Centre Rene Gauducheau, Saint-Herblain
  - Clinique Mutualiste de l'Estuaire - Centre d'oncologie, Saint-Nazaire
  - Institut de Cancerologie de la Loire Lucien Neuwirth, Saint-Priest-en-Jarez
  - Institut de Cancerologie Strasbourg Europe (formar Paul Strauss), Strasbourg
  - CHU Toulouse - Hopital Larrey, Toulouse
  - Gustave Roussy, Villejuif
- Germany (5):
  - Charite - Universitaetsmedizin Berlin - Campus Virchow-Klinikum, Berlin
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Universitaetsklinikum Greifswald der Ernst Morizt Arndt Univ. Greifswald AoR, Greifswald
  - Universitaetsklinikum Jena, Jena
  - Onkologie UnterEms, Leer-Papenburg-Emden, Leer
- Greece (4):
  - NIMTS - Veterans Administration Hospital, Athens
  - Athens University - Attikon University General Hospital, Athens
  - Hygeia Hospital, Athens
  - Ioannina University Hospital, Ioannina
- Italy (15):
  - Ospedale Civile Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - Alma Mater Studiorium Universita di Bologna - Loc. Ospedala Sant'Orsolo, Bologna
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia, Brescia
  - Azienda Istituti Ospitalieri di Cremona, Cremona
  - IRCCS Azienda Ospedaliera Universitaria San Martino "IST" Istituto Nazionale per la Ricerca sul Cancro, Genova
  - Azienda Unita Locale Socio-Sanitaria N. 9-Mater Salutis Hospital, Legnago
  - IRCCS - Istituto Neurologico Carlo Besta, Milan
  - Azienda Sanitaria Locale Napoli 1 Centro, Napoli
  - Universita Di Torino - Ospedale S. Luigi Gonzaga, Orbassano
  - IRCCS - Istituto Oncologico Veneto, Padua
  - Istituti Clinici Scientifici Maugeri, Pavia
  - Regina Elena National Cancer Center, Roma
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino - Ospedale Molinette, Torino
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino - Ospedale San Giovanni - Dipartimento Neuroscienze, Torino
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino - Ospedale Sant'Anna, Torino
- Lithuanian Oncology Center-Nat. Cancer Inst, Vilnius, Lithuania
- Netherlands (5):
  - The Netherlands Cancer Institute-Antoni Van Leeuwenhoekziekenhuis, Amsterdam
  - Amsterdam UMC - Locatie AMC, Amsterdam
  - University Medical Center Groningen, Groningen
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Radboud University Medical Center Nijmegen, Nijmegen
- Poland (4):
  - Medical University Of Gdansk, Gdansk
  - Maria S. Curie Memorial Institute-Gliwice Branch, Gliwice
  - The Great Poland Cancer Centre, Poznan
  - Maria Sklodowska-Curie Memorial Cancer Centre, Warsaw
- Portugal (8):
  - Instituto Portugues De Oncologia - Centro De Coimbra, Coimbra
  - Instituto Portugues de Oncologia de Lisboa Francisco Gentil - EPE, Lisbon
  - Hospital CUF Tejo, Lisbon
  - Centro Hospitalar de Lisboa Ocidental- San Francisco Xavier Hospital, Lisbon
  - Hospital CUF Descobertas, Lisbon
  - Centro Hospitalar do Porto- Hospital de Santo Antonio, Porto
  - Instituto Portugues de Oncologia do Porto, Porto
  - Unidade Local de Saúde Gaia e Espinho, Vila Nova de Gaia
- Medisprof Cancer Center srl, Cluj-Napoca, Cluj Napoca, Romania
- Serbia (2):
  - University Clinic Centre Serbia - Pulmonology clinic, Belgrade
  - University Clinical Center of Serbia - Clinic for ENT and MFH, Belgrade
- Slovenia (2):
  - University Clinic Golnik, Golnik
  - University Medical Center Maribor, Maribor
- Spain (17):
  - ICO L'Hospitalet - Hospital Duran i Reynals (Institut Catala D'Oncologia), L'Hospitalet de Llobregat, Barcelona
  - Vall d'Hebron Institut d'Oncologia, Barcelona
  - Hospital Clinic Universitari de Barcelona, Barcelona
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Hospital General Universitario De Elche, Elche
  - ICO Girona - Hospital Doctor Josep Trueta (Institut Catala D'Oncologia), Girona
  - ICO L'Hospitalet- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario QuironSalud, Madrid
  - Hospital Universitario Virgen De La Victoria, Málaga
  - Hospital Clinico Universitario De Valencia, Valencia
  - Hospital Clinico Universitario De Valladolid, Valladolid
  - Hospital Clinico Universitaro De Valladolid, Valladolid
- Switzerland (3):
  - Hirslanden Klinik-Tumor Zentrum Aarau, Aarau
  - Kantonsspital St Gallen, Sankt Gallen
  - UniversitaetsSpital Zurich, Zurich
- United Kingdom (12):
  - Betsi Cadwaladr University Health Board - Glan Clwyd District General Hospital, Bodelwyddan, Denbighshire
  - University Hospitals Birmingham NHS Foundation Trust (UHB) - UHB-Queen Elisabeth Medical Centre, Birmingham
  - Royal Orthopaedics Hospital, NHS Trust, Birmingham
  - Cambridge University Hospital NHS - Addenbrookes Hospital, Cambridge
  - Velindre NHS Trust - Velindre Cancer Centre, Cardiff
  - University Hospitals Coventry and Warwickshire NHS Trust - University Hospital, Coventry
  - NHS Lothian - Western General Hospital, Edinburgh
  - NHS Greater Glasgow and Clyde - Beatson West of Scotland Cancer Centre - Gartnavel General Hospital, Glasgow
  - Hereford County Hospital, Hereford
  - Leeds Teaching Hospitals NHS Trust - St. James's University Hospital, Leeds
  - Royal Free Hospital, London
  - The Christie NHS Foundation Trust, Manchester